CLINICAL TRIAL: NCT03223805
Title: A Randomised Controlled Trial to Determine the Clinical and Cost Effectiveness of the Respiratory Distress Symptom Intervention for People With Lung Cancer
Brief Title: Respiratory Distress Symptom Intervention (RDSI) Trial
Acronym: RDSI-LC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16_CPCR_01
Record Dates: First submitted 2017-07-12; First posted 2017-07-21 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Other): Usual Care
  Interventions: Other: Respiratory Distress Symptom Intervention
- Intervention Arm (Experimental): Respiratory Distress Symptom Intervention plus Usual Care
  Interventions: Other: Respiratory Distress Symptom Intervention

INTERVENTIONS:
Other: Respiratory Distress Symptom Intervention — The RDSI comprises of four components
  1. Controlled breathing techniques - consists of diaphragmatic breathing exercises and calming techniques practised twice a day and used as needed for episodes of intense breathlessness and/or anxiety
  2. Cough suppression techniques - includes education (capacity for voluntary cough easing, identifying warning signs for cough and replace with modified swallow technique or relaxed throat breath
  3. Acupressure: a small number of acupressure points are taught: L7, L9, LI4 (located on the hand and wrist areas), CV21 and 22 (sternum), and ST36 (knee). Patients can select any of these points in any combination to apply pressure for one-minute at least twice a day for symptom relief
  4. Exercise: Individually-tailored exercise plan, for example, walking incrementally increasing distances in their local environment, incorporating breathing techniques as required

SUMMARY:
This study aims to determine the effects of adding the Respiratory Distress Symptom Intervention (RDSI) to usual care for the self management of the Respiratory Distress Symptom Cluster (breathlessness-cough-fatigue) for patients with lung cancer including mesothelioma.

DETAILED DESCRIPTION:
Lung cancer is responsible for 33,000 deaths each year in the UK and as disease cure is rarely possible, patient management is often aimed at symptom control. Breathlessness, cough and fatigue are common and distressing symptoms occurring in up to 90%, 47-86% and 50-90% of patients respectively. To date, research in relation to this group of symptoms has focussed on breathlessness, cough or fatigue as single symptoms. However, it is likely that ifa patient suffers from one symptom, they also suffer from one or both of the others. Collectively these symptoms are referred to as the Respiratory Distress Symptom Cluster.

Our group has developed a multi-modal Respiratory Distress Symptom Intervention (RDSI) for the self management of breathlessness, cough and fatigue. This study aims to determine the effects of adding the RDSI to usual care for the self-management of the Respiratory Distress Symptom Cluster for patients with lung cancer.

Patients who take part will be assigned to one of two groups; usual care or usual care plus the RDSI.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of lung cancer - primary tumour, secondary tumour or mesothelioma
2. Suffering from refractory breathlessness or cough or fatigue (presence of a minimum of two of the three symptoms), and which is bothersome to the patient (see below)*
3. In the presence of COPD, in stable condition
4. WHO Performance Status 0-2
5. Expected prognosis of at least 3 months
6. 18+ years
7. able to give informed consent

   * Patients will be asked as part of the symptom screening process:

Are you affected in your day to day life by breathlessness? Are you affected in your day to day life by cough? Are you affected in your day to day life by fatigue?

Exclusion Criteria:

1. Patients who are experiencing breathlessness, cough and/or fatigue but do not find these symptoms bothersome are not eligible (see below)*
2. Acute exacerbation** of COPD, or chest infection, within the past 3 weeks, necessitating a change in medication
3. Rapidly worsening breathlessness requiring urgent medical intervention
4. Post chemotherapy and/or radiotherapy to the chest > 2 weeks
5. Surgical treatment for lung cancer > 4 weeks

   * Patients will be asked as part of the symptom screening process:

Are you affected in your day to day life by breathlessness? Are you affected in your day to day life by cough? Are you affected in your day to day life by fatigue?

** An exacerbation is defined as a sustained worsening of the patient's symptoms from their usual stable state which is beyond normal day-to-day variations, and is acute in onset. Commonly reported symptoms are worsening breathlessness, cough, increased sputum production and change in sputum colour. The change in these symptoms often necessitates a change in medication. NICE guidelines 201025. In this trial, patients will only be excluded if a change in medications were required - i.e. steroids or antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Breathlessness | 12 weeks
  Dyspnoea-12
  Dyspnoea-12(D-12)27. Dyspnoea-12: is the primary outcome for breathlessness. It provides an assessment of total breathlessness severity that incorporates its physical discomfort and emotional consequences. It has been validated in a range of respiratory conditions including lung cancer (unpublished data).
Cough | 12 weeks
  The Manchester Cough in Lung Cancer scale. This is a patient self-report consisting of 10 items. This is the only lung cancer specific scale available for the assessment of cough30. Evidence of MCLC reliability and validity has been further reported in intrathoracic malignancy (unpublished PhD data).
Fatigue | 12 weeks
  The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) This is a 13-item standalone scale with good psychometric properties and established minimally important difference. It is commonly used for the assessment of fatigue in lung cancer with good psychometric properties.

SECONDARY OUTCOMES:
NRS Ability to cope with symptoms. | 12 weeks
  Consists of 3 items, breathlessness, cough and fatigue, each on a NRS ranging from 0 (not able to cope at all) to 10 (completely able to cope).
Mood state - Hospital Anxiety & Depression Scale (HADS) | 12 weeks
  This is a 14-item scale assessing anxiety with 7 items and depression with a further 7 items. Each item is answered on a 4-point scale (0-3). Scores on each sub-scale thus range between 0 (no symptoms) and 21 (numerous and severe symptoms). Higher scores are indicative of more anxiety and depression, scores below 8 are considered to be in the normal range, 8-10 are borderline, and scores above 11 indicates a disorder of relevant mood
EQ-5D-5L | 12 weeks
  EQ-5D is a standardised instrument for use as a measure of health outcome. It is applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys. The EuroQoL 5-level version (EQ-5D-5L) will be assessed to provide a preference based measure of health-related quality-of-life which will enable us to calculate a quality adjusted life-year for use in the cost-effectiveness analysis.
Health care utilisation | 12 weeks
  Assessment of resource use will be assessed via patient-recall using a standardised instrument at baseline (previous 4 weeks), week 4 and week 12. Utilisation of resource being measured include: planned hospital or hospice overnight stays, planned hospital out-patient visits, hospital emergency visits, hospital admissions (days/nights), GP and other community service visits (community nurse, walk-in centre, occupational therapist, care worker, home help, social worker).

OTHER OUTCOMES:
Carer outcome measures. Quality of Life (Caregiver Quality of Life Index-Cancer). | 12 weeks
  This is a 35-item scale evaluating the quality of life of those caring for cancer patients and the impact of caregiving on carers' life.
Carer outcome measures. Mood state (Hospital Anxiety & Depression Scale). | 12 weeks
  This is a 14-item scale assessing anxiety with 7 items and depression with a further 7 items. Each item is answered on a 4-point scale (0-3). Scores on each sub-scale thus range between 0 (no symptoms) and 21 (numerous and severe symptoms). Higher scores are indicative of more anxiety and depression, scores below 8 are considered to be in the normal range, 8-10 are borderline, and scores above 11 indicates a disorder of relevant mood.
Carer outcome measures. Fatigue (FACIT-F) | 12 weeks
  The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F )31 This is a 13-item standalone scale with good psychometric properties and established minimally important difference. It is commonly used for the assessment of fatigue in lung cancer with good psychometric properties.

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - University Hospital South Manchester, Manchester, Greater Manchester
  - Heartlands Hospital, Heart of England NHS Foundation Trust, Birmingham
  - Castle Hill Hospital, Hull and East Yorkshire Hospitals NHS Foundation Trust, Cottingham
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - The Clatterbridge Cancer Centre NHS Foundation Tust, Metropolitan Borough of Wirral
  - Scarborough General Hospital, York Teaching Hospital NHS Foundation Trust, Scarborough

REFERENCES:
- [Derived] Yorke J, Johnson MJ, Punnett G, Smith J, Blackhall F, Lloyd Williams M, Mackereth P, Haines J, Ryder D, Krishan A, Davies L, Khan A, Molassiotis A. Respiratory distress symptom intervention for non-pharmacological management of the lung cancer breathlessness-cough-fatigue symptom cluster: randomised controlled trial. BMJ Support Palliat Care. 2024 Jan 8;13(e3):e1181-e1190. doi: 10.1136/spcare-2022-003924. PMID 36283797